CLINICAL TRIAL: NCT05072067
Title: EFFICACY OF THE SLEEVE GASTROPLASTY WITH THE ENDOSCOPIC SYSTEM OVERSTICH SX ON WEIGHT LOSS AND REDUCTION OF CO-MORBIDITY FOR OBESE PATIENTS
Acronym: SLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Trocadéro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A01562-39
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OBESE PATIENT (Experimental): OverStitch™ Sx with a Single channel endoscop CO2 Insufflation, patient on decubitus dorsal, with intubate 3 to 7 sutures, from the antral ogiv to the cardia are done
  Interventions: Procedure: the sleeve gastroplasty with the endoscopic system Overstich SX

INTERVENTIONS:
Procedure: the sleeve gastroplasty with the endoscopic system Overstich SX — the sleeve gastroplasty with the endoscopic system Overstich SX

SUMMARY:
The OverStitch ™ Sx System (Apollo Endosurgery Inc., Austin, Tx, Usa) is a new generation of endoscopic suturing device. It is inserted into an endoscope allowing the approximation of Luc Karsentys soft tissue by placement of sutures. It is as effective a suture system as a surgical system. The OverStitch ™ Sx allows suturing in the upper and lower GI with a flexible single channel endoscope. Previously, the ™ Overstich was only compatible with an Olympus dual channel endoscope.

Thus, a wide range of interventions are possible, including gastric endoplastic sleeve (ESG), RYGB revision, anastomotic fistula repair and / or sleeve revision. In each of these indications, the OverStitch (OverStitch) ™ system has shown its effectiveness and safety.

The OverStitch Endoscopic ™ Suture System allows the entire digestive wall to be sutured through a flexible endoscope. Thus, a wide range of interventions are possible, including gastric pocket repair after gastric bypass surgery, anastomotic fistula repair, endoscopic treatment of digestive perforation, and endoscopic sleeve surgery. In each of these indications, the OverStitch system has demonstrated its effectiveness and safety. But this technique is recent, especially in France. In addition, no data has yet been released regarding the new Overstitch ™ Sx device compatible with all single channel endoscopes.

An observational study including patients in French centers that are experts in therapeutic endoscopy seems essential to us to better assess this new device and this new technique in practice

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18, male or female
* Patient with obesity with a BMI> 30 or BMI> 40 (if surgery contraindicated or refused by the patient)
* Patient with a weight gain after sleeve gastroplasty or sleeve gastrectomy
* Informed and written consent of the patient obtained
* Complete clinical examination
* Lack of participation in another clinical study
* Patient able to follow, understand the study and answer the questionnaire

Exclusion Criteria:

* Haemorrhagic disease, haemostasis and coagulation disorder and platelets <60000 / mm3).
* Breastfeeding women
* Toxicomany, alcoolism
* Patient known for gastric lesion requiring surveillance or familial history of gastric neoplasia
* Hiatus hernia> 4 cm high

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
For the endoscopic sleeve: by the rate of patients with a percentage of total weight lost | 6 MONTHS
For the endoscopic sleeve: by the rate of patients with a percentage of total weight lost | 12 MONTHS

SECONDARY OUTCOMES:
Evaluation of safety Immediate morbidity | DAY 1
For sleeve revision, by the rate of patients with a percentage of total weight lost | 6 MONTHS
For sleeve revision, by the rate of patients with a percentage of total weight lost | 12 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Du Trocadero, Paris, France

IPD SHARING:
Plan to Share IPD: No